CLINICAL TRIAL: NCT02592057
Title: A Multicenter, Prospective, Observational, Post Marketing Surveillance Study to Evaluate the Safety and Efficacy of Sofosbuvir-based Regimens in Clinical Practice for the Treatment of Patients With Chronic Hepatitis C Virus Infection in India
Brief Title: Safety and Efficacy of Sofosbuvir-based Regimens in Clinical Practice for the Treatment of Chronic Hepatitis C Virus Infection in India
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-334-1775
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SOF-based regimens: Adults with chronic HCV infection in India who are being treated with a SOF-based treatment regimen as per the approved prescribing information.
  Interventions: Drug: SOF

INTERVENTIONS:
Drug: SOF — SOF tablets administered orally once daily based on approved prescribing information
  Other Names: Sovaldi ®; GS-7977

SUMMARY:
This study will evaluate the safety and efficacy of sofosbuvir (SOF)-based regimens administered as per the approved prescribing information in adults with chronic hepatitis C virus (HCV) infection treated in routine clinical practice in India.

ELIGIBILITY:
Inclusion Criteria:

* HCV-infected patients living in India
* Treatment with a SOF-based regimen as determined by the patient's treating physician per the approved prescribing information.
* Patients who provide written and signed informed consent prior to initiation of treatment where required.

Exclusion Criteria:

* Concurrent participation in an HCV clinical trial (except trials not testing investigational medicinal products)
* Patients presenting a risk of not being able to be followed (eg, patients planning to move or leave the country in a foreseeable future)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults residing in India aged ≥ 18 years, who are infected with HCV, and for whom the treating physicians in the participating clinics have prescribed a SOF-based regimen as per the approved prescribing information.
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) during treatment and up to 4 weeks after discontinuation of a SOF-based regimen | Up to Posttreatment Week 4

SECONDARY OUTCOMES:
Proportion of participants with sustained virologic response (SVR) 12 weeks after discontinuation of therapy (SVR12) | Posttreatment Week 12
  SVR12 is defined as HCV RNA < the lower limit of quantification (LLOQ) 12 weeks following the last dose of study drug, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (26):
- India (26):
  - Global Hospitals, Hyderabad, Andhra Pradesh
  - A.I.I.M.S., New Delhi, Ansari Nagar
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - Artemis Hospital, Gurgaon, Haryana
  - Manipal Hospital, Bengaluru, Karnataka
  - BGS global Hospitals, Bengaluru, Karnataka
  - Lakeshore Hospital, Kochi, Kerala
  - Midas Institute of Gastro-enterology, Nagpur, Maharashtra
  - S.R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Marudhar Hospital, Jaipur, Rajasthan
  - Global Hospitals & Health City, Chennai, Tamil Nadu
  - VGM Hospital, Coimbatore, Tamil Nadu
  - KGMU Medical College, Lucknow, Uttar Pradesh
  - Postgraduate Institute of Medical Education and Research, Chandigarh, Uttarakhand
  - Institute of Post Graduate Medical Education And Research, Kolkata, West Bengal
  - Sanjivani Superspeciality Hospital Clinical Research Department, Ahmedabad
  - Saviour Hospital, Ahmedabad
  - Sri Ramachandra Medical College and Research, Chennai
  - Aware Global Hospital, Hyderabad
  - M.V. Hospital and Research Centre, Lucknow
  - K. R. M. Hospital & Research Centre, Lucknow
  - Dayanand Medical College & Hospital, Ludhiana
  - BYL Nair Hospital & T N Medical College, Mumbai
  - Sir Ganga Ram Hospital, New Delhi
  - Om Research Center, Om Surgical Center & Maternity Home, Varanasi